CLINICAL TRIAL: NCT05735704
Title: Early Detection and Screening of Hematological Malignancies - SANGUINE
Acronym: SANGUINE
Status: Recruiting | Type: Observational
Sponsor: JaxBio Ltd (Industry)
Collaborators: Tel Aviv University (Other); FORSCHUNGSZENTRUM FUR MEDIZINTECHNIK UND BIOTECHNOLOGIE (Unknown); University Hospital Olomouc (Other); Faculty of Medicine and Dentistry, Palaky University Olomouc (Unknown); Vilnius University Hospital Santaros Klinikos (Other); PREDICTBY RESEARCH AND CONSULTING S.L. (Unknown); National Kapodistrian University of Athens (Unknown); Tel-Aviv Sourasky Medical Center (Other Government); UAB ORIENTOS (Unknown); EUROPEAN CANCER ORGANISATION (Unknown); Predict * By (Unknown); JaxBio Technologies (Unknown)
Responsible Party: Sponsor
Other Study IDs: SANGUINE
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hematologic Malignancy
Keywords: Multiple myeloma; Pre-MM conditions; Hodgkin Lymphoma; Non-Hodgkin aggressive lymphoma; High Grade Lymphoma; Follicular Lymphoma; Marginal zone lymphoma; Acute Myeloid Leukemia; Myelodysplastic syndrome; Diffuse large B cell lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Large B-Cell, Diffuse | interventions — Blood Specimen Collection; Diagnostic Techniques and Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and bone marrow samples are collected and stored for 15 years from the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with Hematological Malignancies - Discovery stage: The first stage (discovery phase) will include at least 30 patients from each of the following groups: MM, pre-MM conditions (SMM and MGUS), HL, aggressive NHL (DLBCL, FL, MZL, AML, MDS.
  NOTE: Patients diagnosed with DLBCL that is transformed from FL or MZL, and patients diagnosed with AML secondary to MDS or MPN, that were treated for their primary disease (FL/MZL/MDS/MPN) prior to study enrollment, are eligible. Patients with a diagnosis of acute promyelocytic leukemia (APL) will not be included.
  For patients, it is expected, after signing the informed consent, that the serial samplings will be performed during the disease follow-up according to the standard clinical practice and/or recommended schedule and disease assessment plan.
  Interventions: Diagnostic Test: Blood sampling for HemaChip screening/diagnostic testing
- Patients with Hematological Malignancies - Second stage: In the second stage, at least 250 patients with MM, 250 patients with NHL, and at least 100 patients with each of the remaining hematological malignancies mentioned above will be tested. Out of these patients, AML, lymphoma, and MM patients will be followed up on at the clinical sites. Periodic sampling will be defined according to disease type and progression rate. Blood and plasma samples will be stored at clinical sites until relapse diagnosis. At this stage, blood samples will be analyzed retrospectively on the HemaChip. The screening, enrollment, and sample collection can begin in the first stage of the trial, to allow a maximum follow-up period for at-risk subjects as part of the study and to meet the recruitment goals.
  Interventions: Diagnostic Test: Blood sampling for HemaChip screening/diagnostic testing
- Subjects at risk of developing MM / lymphoproliferative disorder - Third stage: The last stage consists of screening of a larger group of subjects at risk of developing MM / lymphoproliferative disorder. This stage will include 400 elderly patients (>65 years old) and 500 first-degree relatives of patients (and in particular siblings). The screening, enrollment, and sample collection can begin in the first stage of the trial, in order to meet the recruitment goals.
  Interventions: Diagnostic Test: Blood sampling for HemaChip screening/diagnostic testing
- Control subjects with no malignant disease- Discovery stage: Control subjects with no malignant disease that serve as controls are expected to donate blood a single time. Following this donation, their participation will end.
  Interventions: Diagnostic Test: Blood sampling for HemaChip screening/diagnostic testing

INTERVENTIONS:
Diagnostic Test: Blood sampling for HemaChip screening/diagnostic testing — Classification of a broad spectrum of blood cancers based on detection of epigenetic biomarkers from genomic DNA, cell-free (cf) DNA, exosomal DNA, RNA, and non-coding RNA. The identified biomarkers will include proteins, metabolites, and other characteristic biomolecules.
  Year 1: During the discovery phase, all tests will be conducted by JaxBio and TAU with the aid of technical service providers. At this stage, microarray measurements will be performed on a commercial platform that will be purchased from Agilent / Illumina. All reagents needed for the test will be either purchased or produced in-house.
  Years 2-3: Throughout the second phase of the project, a custom-targeted microarray, HemaChip will be developed and used for all tests. The HemaChip and custom reagents will be distributed to partners' labs and all tests will be conducted at the clinical sites. Additional validation tests will be conducted by JaxBio and TAU, as needed.
  Other Names: HemaChip

SUMMARY:
This is a multicenter, open-label, non-interventional controlled study to identify and characterize the epigenetic signatures for a set of hematological malignancies: Multiple myeloma (MM), pre-MM conditions [smoldering MM (SMM) and monoclonal gammopathy of undetermined significance (MGUS)], Hodgkin lymphoma (HL), diffuse large B cell lymphoma (DLBCL), Follicular lymphoma (FL), Marginal Zone lymphomas (MZL), acute myeloid leukemia (AML)*, myelodysplastic syndrome (MDS), subjects at risk and control subjects with no malignant disease.

*Patients with a diagnosis of acute promyelocytic leukemia (APL) are not included

DETAILED DESCRIPTION:
Subjects will be screened for eligibility and then, after signing an Informed Consent Form, the first peripheral blood sample will be obtained.

Periodical blood samples will be obtained from the participants. Relapse patients will have their retrospective blood samples analyzed to identify early signs of disease.

The first stage (discovery phase) will include at least 30 patients from each of the following groups: MM, pre-MM conditions (SMM and MGUS), HL, DLBCL, FL, MZL, AML, MDS, and control subjects with no malignant disease.

In the second stage, at least 250 patients with MM 250 patients with NHL, at least 100 patients with each of the remaining hematological malignancies mentioned above, and control subjects with no malignant disease will be tested. Out of these patients, AML, lymphoma and MM patients will be followed up at the clinical sites. Periodic sampling will be defined according to disease type and progression rate. Blood and plasma samples will be stored in the clinical sites until relapse diagnosis. At this stage, blood samples will be analyzed retrospectively on the HemaChip. The screening, enrollment, and blood collection can begin in the first stage of the trial, to allow a maximum follow-up period, as part of the study, and to meet the recruitment goals.

The last stage consists of the screening of a larger group of subjects at risk of developing MM / lymphoproliferative disorder. This stage will include 400 elderly patients (>65 years old) and 500 first-degree relatives of patients (and in particular siblings). The screening, enrollment, and sample collection can begin in the first stage of the trial, to allow a maximum period for at-risk subjects cohort to meet the recruitment goals.

In all stages, the age and sex-matched subgroups will be considered and matched.

During the follow-up period, demographic and baseline parameters including sex, age, race, height and weight, medical history, smoking status, details of initial diagnosis and treatment history, concomitant medications as well as adverse events (AEs) of special interest, (serious) AEs related to study procedures, treatment for the disease, disease response and survival status will be collected (as applicable).

ELIGIBILITY:
Inclusion Criteria:

General criteria for all study populations:

1. Male and female subjects ≥18 years of age
2. Ability to understand and willingness to sign a written informed consent document.

For Patients with hematological malignancies:

1. Patients who have been diagnosed, have measurable disease, and/or are being monitored/followed up due to one of the following conditions: MM, pre-MM conditions (SMM and MGUS), HL, DLBCL, FL, MZL, AML, MDS that did not yet undergo any treatment.

NOTE:

Patients diagnosed with DLBCL that is transformed from FL or MZL, and patients diagnosed with AML secondary to MDS or MPN, who were treated for their primary disease (FL/MZL/MDS/MPN) before study enrollment, are eligible.

For subjects at risk for developing the investigated hematological malignancies:

1. First-degree relatives; AND /OR
2. Elderly subjects ≥ 65 years of age.

Exclusion Criteria:

1. Patients/subjects with current co-diagnosis of another type of cancer;
2. Patients/subjects with a known active or prior cancer (other than defined as study population), occurring within the last 2 years (even if considered to be in complete remission). Patients/subjects with non- melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection;
3. Patients with a diagnosis of acute promyelocytic leukemia (APL)
4. Patients/subjects with active inflammatory autoimmune disease that requires treatment with immunosuppressive/ immunomodulation agents;
5. Patients/subjects with known human immunodeficiency virus (HIV) positive;
6. Patients/subjects with known active Hepatitis A/B/C or past hepatitis C;
7. Subjects that are likely to be noncompliant with the protocol, or felt to be unsuitable by the investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — older then 18 year old
Study Population: Adult subjects with hematological malignancies: Multiple myeloma (MM), pre-MM conditions [smoldering MM (SMM) and monoclonal gammopathy of undetermined significance (MGUS)], Hodgkin lymphoma (HL), non-Hodgkin aggressive lymphoma NHL [diffuse large B cell lymphoma (DLBCL), FL, MZL, acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), subjects at risk and control subjects with no malignant disease.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker discovery | 36 month
  define a set of differential epigenetic biomarkers that uniquely identify the following conditions: MM, pre-MM conditions (SMM and MGUS), HL, aggressive NHL (DLBCL, HGL, FL and MZL transformed to large cell lymphoma), FL, MZL, de novo AML, secondary AML, MDS and healthy subjects.
Validation of Hemachip | 36 month
  Validating the discovery platform (HemaChip) as a diagnostic tool for various blood cancers.
Early detection for hematological malignancies | 36 month
  Towards early detection - Patients, at risk of relapse tested periodically to evaluate early detection capability of the HemaChip.
population screening for hematological malignancies | 36 month
  Towards population screening - evaluate the sensitivity and specificity for screening in populations at risk for developing the investigated cancers: (i) elderly (>65 years old) at high risk to develop MM; (ii) first degree relatives of the conditions described above.

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Prof. Ebenstein, PhD, Study Chair — Tel Aviv University
Locations (4):
- Fakultni Nemocnice Olomouc (Fnol), Olomouc, Czechia
- National and Kapodistrian University of Athens (NKUA), Athens, Greece
- Tel-Aviv Sourasky Medical Center (TASMC), Tel Aviv, Israel
- Vilnus University Hospital Santaros Klinikos (VULSK), Vilnius, Lithuania